CLINICAL TRIAL: NCT04256785
Title: Efficacy and Tolerability of the Probiotic VSL#3 for the Treatment of Patients With Fibromyalgia and Associated Gastrointestinal Symptomatology: a Randomized, Double-blind Clinical Trial
Brief Title: Probiotic VSL#3 for the Treatment of Gastrointestinal Symptoms Associated to Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elena Pita Calandre (Other)
Collaborators: Actial Farmaceutica S.r.l. (Industry); Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Elena Pita Calandre, professor, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMS-VSL3-19
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Fibromyalgia; Gastrointestinal Disease
Keywords: probiotic; efficacy; tolerability
MeSH Terms: conditions — Fibromyalgia; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSL#3 (Experimental): probiotic VSL#3, 2 sachets b.i.d for 3 months
  Interventions: Dietary Supplement: VSL#3
- placebo (Placebo Comparator): matched placebo, 2 sachets b.i.d for 3 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — sachets containing probiotic
  Arms: VSL#3
Dietary Supplement: Placebo — sachets containing placebo
  Arms: placebo

SUMMARY:
The study evaluated the efficacy and tolerability of probiotic VSL#3 for the treatment of gastrointestinal symptoms in patients with fibromyalgia; 50% of the participants received probiotic and the remaining 50% received matching placebo in a double-blind, randomized design.The treatment was administered during a 12-week period and the participants were followed for an additional 12-week period in order to follow the evolution after treatment.

DETAILED DESCRIPTION:
Many patients with fibromyalgia experience associated gastrointestinal symptomatology such as abdominal pain, abdominal bloating, meteorism, diarrhea and/or constipation. To date there is not any specific treatment for these symptoms that markedly impair the quality of life of these subjects. This trial intended to investigate if the addition of a polymicrobial probiotic product, which has shown efficacy in patients with irritable bowel syndrome, was also be useful to ameliorate the gastrointestinal symptomatology of patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed of fibromyalagia
* experiencing at least 3 chronic gastrointestinal symptoms
* signed informed consent to participate
* accept to not change previously prescribed treatment during study duration

Exclusion Criteria:

* mental illness excepting depression
* severe organic disease
* additional gastrointestinal disease excepting irritable bowel syndrome
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena P. Calandre, M.D., Principal Investigator — Universidad de Granada
Locations (1):
- Instituto de Neurociencias "Federico Oloriz", Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after study completion
Access Criteria: Data access requests will be reviewed by study sponsor and P.I.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VSL#3 | Placebo
Started | 54 | 56
Completed | 26 | 31
Not Completed | 28 | 25
Not completed — Adverse Event | 8 | 6
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 7 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Surgery or quarantined due to Covid-19 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VSL#3 | Placebo | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7.5) | 55.5 (8.6) | 55.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 107
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 56 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight (Kg) [Mean (Standard Deviation); unit: kgs] | 73.3 (17.7) | 71.2 (13.4) | 72.2 (15.6)
Fibromyalgia diagnosis - Widespread Pain Index (WPI) total score [Mean (Standard Deviation); unit: scores on a scale] — The WPI assesses presence of pain in 19 designated body locations over the past 7-days. Each location is equal to a score of 1. Items are summed to yield a total score, with higher scores indicating greater widespread pain.
  scores on a scale | 15.9 (3.0) | 16.5 (2.6) | 16.2 (2.8)
Fibromyalgia diagnosis - Symptom Severity Score [Mean (Standard Deviation); unit: scores on a scale] — The SSS is a scale that evaluates the presence and severity of associated symptoms, excluding pain, in patients with fibromyalgia. The SSS total score is calculated by summing the 0-3 scores of somatic symptoms, waking unrefreshed, cognition, and fatigue into a 0-12 scale. Higher scores indicate more associated symptoms of higher severity.
  scores on a scale | 9.3 (2.0) | 9.7 (1.7) | 9.5 (1.9)
Fibromyalgia diagnosis - Fibromyalgia Score [Mean (Standard Deviation); unit: scores on a scale] — The FS score is the sum of WPI and SSS. The total score ranges from 0 to 31 points. Higher scores indicate higher fibromyalgia severity scores.
  scores on a scale | 25.3 (4.3) | 26.2 (3.5) | 25.7 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change, From Baseline to Endpoint (12 Weeks) in the Composite Score of Abdominal Pain, Abdominal Bloating and Metheorism Each One Measured in a 0-10 Visual Analog Scale
Description: Visual analogue scales are frequently used to evaluate subjective symptoms; they range from 0 (no symptom at all) to 10 (worst possible intensity of the symptom) points. In the present case the three most frequent abdominal symptoms reported by patients with fibromyalgia have been selected to compose the primary outcome variable. Total symptoms range was 0 to 30 points. Change = (week 12 score - baseline score)
Time Frame: baseline and twelve weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- VSL#3: probiotic VSL#3, 2 sachets b.i.d for 3 months
  VSL#3: sachets containing probiotic
  54 subjects
- Placebo: matched placebo, 2 sachets b.i.d for 3 months
  Placebo: sachets containing placebo
  56 subjects
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | -6.5 (9.5) | -5.4 (6.6)

2. Secondary Outcome: Change, From Baseline to Endpoint (12 Weeks) in the Total Score of the Fibromyalgia Impact Questionnaire Revised (FIQR)
Description: The FIQR is a self-reported, validated questionnaire that evaluates the severity of fibromyalgia symptomatology in a scale ranging from 0 to 100 points; the higher the score, the worse the severity of the disease. Change = (week 12 score - baseline score)
Time Frame: baseline and twelve weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | -7.2 (12.5) | -12.5 (14.1)

3. Secondary Outcome: Change, From Baseline to Endpoint (12 Weeks) in the Total Score of the Insomnia Severity Inventory (ISI)
Description: The ISI is a self-reported, validated questionnaire that measures the severity of sleep disturbances in a scale ranging from 0 to 28 points: higher scores indicate more severe sleep disturbance
Time Frame: baseline and twelve weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | -1.7 (5.9) | -1.2 (4.0)

4. Secondary Outcome: Change, From Baseline to Endpoint (12 Weeks) in the Total Score of the Patient Health Questionnaire (PHQ-9)
Description: PHQ-9 is a self-reported, validated questionnaire that measures the severity of depression in a scale ranging from 0 to 27 points; higher scores indicate more severe depression. Change = (week 12 score - baseline score)
Time Frame: baseline and twelve weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | -2.2 (7.2) | -2.5 (4.2)

5. Secondary Outcome: Change, From Baseline to Endpoint (12 Weeks) in the Short-Form Health Survey SF-36 PCS
Description: The SF-36 is a self-reported, validated questionnaire evaluating the general health quality in a scale ranging from 0 to 100 points; it evaluates 8 heath domains that yield two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Higher scores indicate better general health quality. Change = (week 12 score - baseline score).
Time Frame: baseline and twelve weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | 4.5 (8.0) | 2.2 (6.3)

6. Secondary Outcome: Change, From Baseline to Endpoint (12 Weeks) in the Short-Form Health Survey SF-36 MCS
Description: as for outcome 5
Time Frame: baseline and 12 weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | 0.8 (12.4) | 1.9 (12.2)

7. Secondary Outcome: Number of Patients Considered as Responders to Treatment
Description: Patients that showed at least a a 30% reduction in the score of the primary variable, i.e. the composite ccore of abdominal pain, abdominal bloating and metheorism each one measured in a 0-10 Visual Analog Scale, were considered as responders to treatment.
Time Frame: Baseline and 12 weeks after treatment
Population: Intent to Treat Population (all patients with at least a post-baseline evaluation)
Measure: Number; unit: participants
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 53 | 53
participants | 27 | 22

8. Secondary Outcome: Change From Week 12 to Week 16 (Follow-up Period) in the Composite Score of Abdominal Pain, Bloating and Metheorism Among Responders After Discontinuing the Study Treatment
Description: Visual analogue scales are frequently used to evaluate subjective symptoms; they range from 0 (no symptom at all) to 10 (worst possible intensity of the symptom) points. In the present case the three most frequent abdominal symptoms reported by patients with fibromyalgia have been selected to compose the primary outcome variable. Total symptoms range was 0 to 30 points. Change = (week 16 score - week 12 score)
Time Frame: Week 12 to week 16
Population: Patients considered as responders to treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 27 | 22
units on a scale | 2.0 (5.2) | 1.7 (4.2)

9. Secondary Outcome: Change From Week 12 to Week 20 (Follow-up Period) in the Composite Score of Abdominal Pain, Bloating and Metheorism Among Responders After Discontinuing the Study Treatment
Description: Visual analogue scales are frequently used to evaluate subjective symptoms; they range from 0 (no symptom at all) to 10 (worst possible intensity of the symptom) points. In the present case the three most frequent abdominal symptoms reported by patients with fibromyalgia have been selected to compose the primary outcome variable. Total symptoms range was 0 to 30 points. Change = (week 20 score - week 12 score)
Time Frame: Week 12 to week 20
Population: Patients considered as responders to treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 27 | 22
units on a scale | 1.0 (3.7) | 3.4 (5.4)

10. Secondary Outcome: Change From Week 12 to Week 24 (Follow-up Period) in the Composite Score of Abdominal Pain, Bloating and Metheorism Among Responders After Discontinuing the Study Treatment
Description: Visual analogue scales are frequently used to evaluate subjective symptoms; they range from 0 (no symptom at all) to 10 (worst possible intensity of the symptom) points. In the present case the three most frequent abdominal symptoms reported by patients with fibromyalgia have been selected to compose the primary outcome variable. Total symptoms range was 0 to 30 points. Change = (week 24 score - week 12 score)
Time Frame: Week 12 to week 24
Population: Patients considered as responders to treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VSL#3 | Placebo
Number analyzed (Participants) | 27 | 22
units on a scale | 1.3 (3.6) | 4.1 (5.5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were collected at each visit during the 12 weeks treatment period.
Arm/Group | VSL#3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 20/54 | 19/56
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VSL#3 (N=54) | Placebo (N=56)
abdominal distension (Gastrointestinal disorders) | 5 (5) | 1 (1)
flatulence (Gastrointestinal disorders) | 5 (5) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Disease worsening (General disorders) | 2 (2) | 0 (0)
Dispepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Swelling (General disorders) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
The high number of patients in both groups that prematurely withdrew from the study for reasons unrelated with treatment tolerability and/or efficacy, hinders the trials capacity to accurately evaluate efficacy of the studied probiotic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT04256785/Prot_SAP_000.pdf